CLINICAL TRIAL: NCT06299475
Title: Structured Online Contraceptive Counseling At Emergency Contraception Pharmacy Provision - a Cluster Randomized Crossover Trial - (The LOWEC Trial)
Brief Title: Structured Online Contraceptive Counseling (LOWE Trial) At Emergency Contraception (EC) Pharmacy Provision LOWE+EC=LOWEC
Acronym: LOWEC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: the Swedish Pharmacy Association (Unknown)
Responsible Party: Principal Investigator, Karin Emtell Iwarsson, Registered nurse-midwife, PhD, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-06755-01
Record Dates: First submitted 2024-01-25; First posted 2024-03-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Contraception
Keywords: eHealth; Emergency Contraception; Over-the-counter

STUDY DESIGN:
Intervention Model Description: A cluster randomized crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online counseling and invitation (Experimental): Participants receive structured online contraceptive counseling and an online invitation to a clinic for contraceptive provision
  Interventions: Other: Online counseling and invitation
- Control (No Intervention): Participants receive standard praxis i.e. no contraceptive counseling or online invitation

INTERVENTIONS:
Other: Online counseling and invitation — Online counseling - An educational video including contraceptive models, four key questions and an effectiveness chart (the LOWE intervention material).
  Invitation to a clinic - access by weblinks to a regional or national website
  Arms: Online counseling and invitation

SUMMARY:
To increase sexual and reproductive health and rights through the improvement of contraceptive counseling and easy access to service and, thus, women's use of effective contraceptives after purchase of an emergency contraceptive pill (ECP).

DETAILED DESCRIPTION:
This pragmatic cluster randomised cross-over controlled trial aims to determine whether the composite intervention of online contraceptive counseling at the time of a pharmacy provision of emergency contraceptive pill (ECP), plus an invitation to a sexual and reproductive health clinic, will result in increased use of subsequent effective contraception (hormonal or intrauterine) compared with standard care.

The study will be conducted at approximately 30 pharmacies in the Stockholm Region. Clients who will buy an ECP (without prescription) at one of these pharmacies will be invited by posters and pharmacy personnel to participate in the study. By scanning a quick response (QR) code they will receive more information about the study. Eligible women who choose to participate in the study and give their consent will be allocated to intervention or control group depending on the visited pharmacy's allocation.

Participants at the intervention pharmacies will receive an intervention package with online structured contraceptive counseling followed by an online invitation to a clinic for contraceptive provision. While participants at the control pharmacies will purchase the ECP without any further guidance. The order in which the pharmacies will provide the intervention or control will be randomly assigned at a ratio 1:1 by an independent statistician. The recruitment will halter for an intervening period of at least two weeks when the pharmacies switch to the new group depending on their first allocation (cross-over).

An online baseline questionnaire and follow-up questionnaires will be collected at 1 and 12 months following the ECP provision for participants both from intervention and control pharmacies.

The randomized controlled trial will be conducted together with a process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Women >/=15 years visiting a pharmacy to buy ECP for her own use
* Has a smartphone with an electronic identification and ability to scan a QR code
* Ability to read Swedish or English
* Willing and able to provide informed consent
* Willing to participate in the follow-up

Exclusion Criteria:

* Ongoing pregnancy

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Use of effective contraception | at 1 month follow-up from the pharmacy visit
  Participant´s self-reported use in a digital questionnaire of regular effective contraception (hormonal or intrauterine)

SECONDARY OUTCOMES:
Contraceptive use | within 12 months follow-up
  Contraceptive use, including long-acting reversible contraception (LARC) (self-reported use in a digital questionnaire)
Incidence of pregnancy and abortion | within 12 months follow-up
  Pregnancy and abortion (self-reported use in a digital questionnaire or scrutinized medical record, if lost to follow-up)
Satisfaction with the intervention | At 1 month follow-up from the pharmacy visit
  Participants' satisfaction with the intervention package (self-reported use in a digital questionnaire) Assessed as: very satisfied, satisfied, neither nor, dissatisfied, very dissatisfied
Contraceptive use, pregnancy, abortion and satisfaction in vulnerable groups | within 12 months follow-up
  Contraceptive use, pregnancy, abortion and satisfaction in vulnerable groups such as youths and migrants, compared to non-migrants and older participants (self-reported use in a digital questionnaire or scrutinized medical record, if lost to follow-up)
Process evaluation | within 12 months follow-up
  How context affects the implementation and outcomes among participants and pharmacy personnel (individual interviews)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Emtell Iwarsson, PhD, Principal Investigator — WHO-centre, Karolinska Institutet, Sweden
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Some unidentified participant data can be shared on request
Time Frame: 2025 - 2027
Access Criteria: Some unidentified participant data can be shared on request